CLINICAL TRIAL: NCT07293728
Title: A Randomized Feasibility Trial Comparing Drospirenone and Norethindrone for Postpartum Hypertension Management in Preeclampsia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Julia Tasset, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00028768
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Preeclampsia
Keywords: Postpartum Hypertension Management
MeSH Terms: conditions — Hypertension; Pre-Eclampsia | interventions — Norethindrone; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Postpartum Norethindrone (Active Comparator): Norethindrone is a well-established progestin-only contraceptive that is considered standard of care for postpartum contraception, particularly in breastfeeding individuals. Norethindrone serves as the comparator arm representing the current standard practice for postpartum contraception in individuals with recent hypertensive disorders of pregnancy.
  Interventions: Drug: Norethindrone 0.35 MG
- Postpartum Drospirenone (Experimental): Drospirenone is a newer progestin-only contraceptive approved by the FDA that exhibits mineralocorticoid receptor activity that has been shown to modestly lower blood pressure in addition to serve as contraception. Drospirenone represents a novel therapeutic option that may offer superior blood pressure outcomes in postpartum individuals with hypertensive disorders unlike other progestin-only contraceptives.
  Interventions: Drug: Drospirenone

INTERVENTIONS:
Drug: Norethindrone 0.35 MG — 1 tablet (0.35 mg) once daily, taken at the same time each day between hospital discharge following delivery until 6 weeks postpartum.
  Arms: Postpartum Norethindrone
Drug: Drospirenone — 1 tablet (4 mg) once daily for 24 days, followed by 4 inactive tablets. Repeated from hospital discharge following delivery until 6 weeks postpartum.
  Arms: Postpartum Drospirenone

SUMMARY:
This is an open-label, randomized feasibility trial in which patients admitted to Oregon Health & Science University (OHSU) after a pregnancy complicated by preeclampsia who are considering a progestin-only pill contraception postpartum will be randomized to norethindrone or drospirenone for 6 weeks following hospital discharge.

DETAILED DESCRIPTION:
In this open-label, randomized, feasibility trial, we will recruit participants admitted to OHSU after a pregnancy complicated preeclampsia (diagnosed antepartum or postpartum). All patients admitted after a birth are offered contraception as a routine part of clinical care; only prospective participants who are undecided in their birth control method or who are considering a progestin-only pill contraception will be approached for inclusion.

Participants who consent for enrollment will be randomized to norethindrone or drospirenone. Prescriptions will be filled by the OHSU research pharmacy and delivered to patients prior to discharge. Participants will then receive weekly emails to report medication adherence, home-measured blood pressures (typical standard of care for preeclampsia), and any interval changes in medication or unscheduled healthcare encounters. Follow up will continue through six weeks, consistent with typical close blood pressure monitoring for postpartum patients with preeclampsia. Participants accessing drospirenone through the study who desire to continue after conclusion will be provided with information for obtaining a prescription from their primary provider as well as manufacturer information to reduce prescription costs (as prior authorization requirements are more common with this medication).

ELIGIBILITY:
Inclusion Criteria:

* Admission to Oregon Health & Science University following a birth (during the same admission)
* A diagnosis of preeclampsia or chronic hypertension with superimposed preeclampsia (with or without severe features)
* Considering use of a progestin-only pill for postpartum contraception

Exclusion Criteria:

* Planned use of a contraceptive method other than a progestin-only pill
* Contraindications to drospirenone or norethindrone
* Inability to monitor blood pressure at home after discharge
* Inability to complete follow-up surveys by email in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Measured weekly for the 6 weeks following delivery.
  Arterial, systolic, and diastolic blood pressure will be compared between norethindrone and drospirenone users. Measured by participants at home and reported in weekly surveys.

SECONDARY OUTCOMES:
Antihypertensive Medications | Collected weekly for the 6 weeks following delivery.
  The proportion of participants requiring up titration or new initiation of antihypertensive medications after discharge from the hospital. Measured by weekly survey.
Follow-Up Visits | Assessed weekly between delivery and 6 weeks postpartum.
  The number of participants requiring unscheduled in-person assessment of blood pressure concerns or readmission to the hospital relating to blood pressure concerns. Will be measured using weekly participant surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Tasset, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time to share individual participant data with other researchers.